CLINICAL TRIAL: NCT00382031
Title: An Open-Labeled Randomized Parallel Group Trial of Zalutumumab, a Human Monoclonal Anti-EGFr Antibody, in Combination With Best Supportive Care (BSC) vs BSC, in Pts With Non-Curable SCCHN Who Have Failed Standard Platinum-Based Chemotherapy
Brief Title: Zalutumumab in Patients With Non-curable Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hx-EGFr-202
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Results first posted 2013-10-15 (Estimated); Last update posted 2013-10-15 (Estimated); Status verified 2013-08

CONDITIONS: Head and Neck Cancer; Squamous Cell Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms, Squamous Cell | interventions — zalutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zalutumumab (Active Comparator): Zalutumumab in combination with Best Supportive Care
  Interventions: Drug: Zalutumumab; Other: Control
- Control (Other): Best Supportive Care
  Interventions: Other: Control

INTERVENTIONS:
Drug: Zalutumumab — Individual dose titration weekly i.v doses
  Other Names: Zalutumumab in combination with Best Supportive Care
  Arms: zalutumumab
Other: Control — Best Supportive Care
  Other Names: Best Supportive Care

SUMMARY:
The purpose of this study is to investigate if zalutumumab in combination with Best Supportive Care (BSC) is superior to BSC in non-curable patients with head and neck cancer

DETAILED DESCRIPTION:
This is an open parallel group trial. Patients will be randomized in a 2:1 manner to receive either treatment with zalutumumab in combination with Best Supportive Care (BSC) or BSC.

Patients randomized to treatment with zalutumumab in combination with BSC will receive weekly infusions with zalutumumab starting with a loading dose (8mg/kg) followed by weekly maintenance doses until disease progression, intercurrent illness preventing further administration, unacceptable toxicity or patient decision. After Visit 2 the patient should be evaluated for presence of skin rash prior to each infusion to allow dose titration.

Individual dose titration until the patient develops grade 2 skin rash will be applied. The maximum dose used in study will be 16 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females age ≥ 18 years
2. Confirmed diagnosis, initially or at relapse, of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx, considered incurable with standard therapy
3. Failure to at least one course of standard platinum-based chemotherapy

Exclusion Criteria:

1. Three or more chemotherapy regimens other than platinum-based chemotherapy
2. Prior treatment with EGFr antibodies and/or EGFr small molecule inhibitors
3. Past or current malignancy other than SCCHN, except for certain other cancer diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2006-11; Primary Completion 2009-12 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (82):
- Belgium (6):
  - University Hospital Antwerp, Antwerp
  - St-Luc University Hospital, Brussels
  - CHNDRF, Charleroi
  - "University Hospital, Ghent
  - University Hospital Leuven, Leuven
  - Cliniques Saint Pierre, Ottignies
- Brazil (13):
  - BioCancer, Belo Horizonte
  - Hospital Erasto Gaertner, Curitiba
  - Centro Goiano de Oncologia, Goiânia
  - Hospital Araújo Jorge, Goiânia
  - Fundação Amaral Carvalho, Jaú
  - CliniOnco, Porto Alegre
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Cepho - Centro de Estudos e pesquisa em Hematologia e Oncologia, Santo André
  - Santo Andre Diag e Tratamentos, Santo André
  - Centro de Oncologia - InRad HCFMUSP, São Paulo
  - Hospital Heliópolis, São Paulo
  - IBCC - Instituto Brasileiro de Combate ao Câncer, São Paulo
  - UNIFESP, São Paulo - SP
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - London Regional Cancer Program, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - BC Cancer Agency, Vancouver, British Colombia
- North-Estonian Regional Hospital, Tallinn, Estonia
- France (5):
  - Hôpital Beaujon- department of medical oncology, Clichy
  - Centre Oscar Lambrette, Lille
  - Centre Antoine Lacassagne, Nice
  - Hôpital Tenon - department of medical oncology, Paris
  - Institut Gustave Roussy, Villejuif
- Hungary (9):
  - Semmelweis University, Budapest
  - Uzsoki Hospital Budapest, Budapest
  - University of Debrecen, Debrecen
  - Petz Aladár, Győr
  - Szabolcs-Szatmar-Bereg County Hospital, Nyíregyháza
  - University of Szeged, Szeged
  - Markusovszky County Hospital, Szombathely
  - Szent Borbála County Hospital Oncology Department, Tatabánya
  - Zala County Hospital, Zalaegerszeg-Pózca
- Lithuania (2):
  - Klaipeda Hospital, Klaipėda
  - Vilnius University, Vilnius
- Poland (9):
  - Beskidzkie Centrum Onkologii, Bielsko-Biala
  - Samodzielny Publiczny Szpital Kiniczny Nr1, Gdansk
  - Katedra i Onkologii Collegium, Krakow
  - Szpital Specjalistyczny im. Rydygiera, Krakow
  - Centrum Onkologii, Lublin
  - Zakład Opieki Zdrowotnej MSWiA z Warmińsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - Centrum Onkologii - Instytut im. M. Curie-Skłodowskiej, Warsaw
  - Dolnoslaskie Centrum Onkologii, Wroclaw
  - Szpital Wojewódzki SP ZOZ, Zielona Góra
- Russia (17):
  - Belgorod Regional Oncology Dispensary, Belgorod
  - Regional Oncology Dispensary, Chelyabinsk
  - Republican Clinical Oncology Dispensary, Izhevsk
  - Kursk Regional Oncology Dispencary, Kursk
  - Kursk Regional Oncology Dispensary, Kursk
  - City Clinincal Oncology Dispensary #1, Moscow
  - Moscow Research Institute of Oncology, Moscow
  - NUZ Semashko Central Clinical Hospital No2 OAO, Moscow
  - Russian Oncology Research Center n.a. Blokhin, Moscow
  - GUZ NO Oncology Dispensary, Nizhiy Novgorod
  - Medical Radiological Research Center, Obninsk
  - St. Petersburg State Medical University, Saint Petersburg
  - Sochi Oncology Center, Sochi
  - Stavropol Regional Clinical Oncology Dispensary, Stavropol
  - Tula Region Oncology Dispensary, Tula
  - GUZ Volgograd Region Clinical Oncology Dispensary No1, Volgograd
  - Voronezh Region Clinical Oncology Dispensary, Voronezh
- Serbia (4):
  - Institute for Oncology and Radiology, Belgrade
  - Military Medical Academy, Belgrade
  - Institute of Oncology Sremska Kamenica, Kamenica
  - Clinic of Maxillofacial Surgery Nis, Niš
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Lund University Hospital, Lund
- United Kingdom (9):
  - Musgrove Park Hospital, Taunton, Somerset
  - Royal Surrey County, Guildford, Surrey
  - Bristol Haematology and Oncology Centre, Bristol
  - The Beatson West of Scotland Centre, Glasgow
  - Royal Marsden Hospital, London
  - Christie Hospital, Manchester
  - Newcastle General Hospital, Newcastle
  - Weston Park Hospital, Sheffield
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Machiels JP, Subramanian S, Ruzsa A, Repassy G, Lifirenko I, Flygare A, Sorensen P, Nielsen T, Lisby S, Clement PM. Zalutumumab plus best supportive care versus best supportive care alone in patients with recurrent or metastatic squamous-cell carcinoma of the head and neck after failure of platinum-based chemotherapy: an open-label, randomised phase 3 trial. Lancet Oncol. 2011 Apr;12(4):333-43. doi: 10.1016/S1470-2045(11)70034-1. Epub 2011 Mar 4. PMID 21377930

RESULTS

PARTICIPANT FLOW:
Groups:
- Zalutumumab: Zalutumumab in combination with Best Supportive Care. Patients received weekly infusions of zalutumumab. After a loading dose of 8 mg/kg the dose was reduced to 4 mg/kg and individual dose titration based on skin rash evaluation was performed.
Period: Overall Study
Arm/Group | Zalutumumab | Control
Started | 191 (Of the 191 randomized patients 189 received at least one infusion of zalutumumab) | 95 (Of the 95 randomized patients 94 attended Visit2.)
Completed | 191 | 95
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) was based on the intent-to-treat principle and thus comprised all randomized patients. The FAS was used for evaluation of all efficacy endpoints and was the primary analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zalutumumab | Control | Total
Number analyzed (Participants) | 191 | 95 | 286
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 161 | 77 | 238
  >=65 years | 30 | 18 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 57 (9) | 57 (9) | 57 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 12 | 34
  Male | 169 | 83 | 252
Region of Enrollment [Number; unit: participants]
  Serbia | 5 | 1 | 6
  Estonia | 3 | 1 | 4
  Spain | 1 | 4 | 5
  Lithuania | 2 | 0 | 2
  Russian Federation | 42 | 22 | 64
  United Kingdom | 22 | 10 | 32
  France | 13 | 3 | 16
  Hungary | 37 | 20 | 57
  Canada | 10 | 8 | 18
  Brazil | 7 | 4 | 11
  Belgium | 31 | 20 | 51
  Poland | 14 | 2 | 16
  Sweden | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: A patient's overall survival was defined as the time from the date of randomization until the date of death from any cause, assessed up to 41 months. Overall survival was censored if the patient was lost to follow-up or refused to continue in the trial.
Time Frame: From randomization until death
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zalutumumab | Control
Number analyzed (Participants) | 191 | 95
months | 6.7 [5.8 to 7.1] | 5.2 [4.1 to 6.4]

2. Secondary Outcome: Objective Tumor Response
Description: Objective tumor response assessed according to Response Evaluation Criteria in Solid Tumours (RECIST v 1.0) J Natl Cancer Inst 2000;92:205-16 assessed by CT/MRI. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the longest diameter of target lesions; Overall Response (OR), CR+PR
Time Frame: From date of randomization until the date of death from any cause, assessed up to 41 months.
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Zalutumumab | Control
Number analyzed (Participants) | 191 | 95
participants
  Complete response | 2 | 0
  Partial response | 10 | 1
  Stable disease | 79 | 25
  Progressive disease | 70 | 38
  Not evaluable | 30 | 31

3. Secondary Outcome: Duration of Response
Description: Duration of response defined as the time from the first date where measurement criteria for complete or partial response (whichever status is recorded first) are met until the first date that death, recurrence or progressive disease is objectively documented.
Time Frame: Time from complete or partial response until death, recurrence or progressive disease, assessed up to 41 months.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Zalutumumab | Control
Number analyzed (Participants) | 12 | 1
month | 5.5 [3.6 to 23.0] | 7.4 [lower limit NA] — CI not available as it was only one patient

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS (defined as the time from randomization until disease progression or death). The progression events were defined by well-documented and verifiable imaging data. In case of censoring, the date of censoring had to be the last time point documenting the status of the patient.
Time Frame: From randomization until disease progression or death, assessed up to 41 months.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Zalutumumab | Control
Number analyzed (Participants) | 191 | 95
weeks | 9.9 [8.7 to 15.0] | 8.4 [8.1 to 9.6]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during weekly visits for patients treated with zalutumumab and visits every fourth week for patients randomized to the control group.
Description: The safety analysis population included all 283 patients who had attended Visit 2.
Arm/Group | Zalutumumab | Control
Serious Adverse Events (participants affected / at risk) | 180/189 | 87/94
Other Adverse Events (participants affected / at risk) | 188/189 | 92/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalutumumab (N=189) | Control (N=94)
General disorders and administration site conditions (General disorders) | 127 (138) | 63 (64)
Disease progression (General disorders) | 118 (118) | 60 (60)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 38 (48) | 22 (27)
Tumour hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 (41) | 14 (17)
Infections and Infestations (Infections and infestations) | 35 (46) | 11 (11)
Pneumonia (Infections and infestations) | 14 (15) | 3 (3)
Gastrointestinal disorders (Gastrointestinal disorders) | 19 (20) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 10 (10) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalutumumab (N=189) | Control (N=94)
General disorders and administration site conditions (General disorders) | 159 (359) | 78 (161)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 174 (355) | 10 (13)
Gastrointestinal disorders (Gastrointestinal disorders) | 102 (298) | 43 (119)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 80 (177) | 33 (51)
Infections and Infestations (Infections and infestations) | 79 (171) | 29 (35)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 77 (150) | 20 (27)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 66 (121) | 26 (44)
Nervous system disorders (Nervous system disorders) | 70 (114) | 22 (38)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 50 (75) | 30 (39)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 46 (78) | 27 (41)
Investigations (Investigations) | 56 (77) | 12 (14)
Vascular disorders (Vascular disorders) | 28 (38) | 7 (9)
Eye disorders (Eye disorders) | 24 (37) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The site and the PI may be required to withhold the publication for up to 90 days. Subject to a reasoned request from the sponsor, the publication may be further delayed for a period up to 6 months from the date of first submission to the sponsor.

The sponsor has the right to require deletion of any trade secret, proprietary, or confidential information supplied by the sponsor to the site or the PI. The sponsor shall not otherwise have the right to censor publications.